CLINICAL TRIAL: NCT00416845
Title: A Randomized, Parallel Group, Double-blind, Placebo Controlled, 14 Days Multiple-dose Treatment to Assess the Pulmonary and Cardiac Pharmacodynamics of FTY720 (0.5 and 1.25 mg) in Healthy Volunteers
Brief Title: Effects of FTY720 on Heart and Lung Functions in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720D2105
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: pharmacodynamic effects, cardiac effects, healthy subjects, synthetic sphingosine 1 phosphate (S1P) receptor modulator; Healthy male and female subjects
MeSH Terms: interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study is designed to assess the effects of two doses of FTY720 on lung (pulmonary) and cardiac (heart) functions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking,(ie. 6 months w/o the use of nicotine or nicotine containing products), male or female subjects.
* Female subjects must be either surgically sterilized (including bilateral tubal ligation) at least 6 months or post-menopausal. Postmenopausal women must have no regular menstrual bleeding for at least 1 year prior to inclusion and menopause will be confirmed by a plasma FSH level of >40 IU/L.
* Male subjects agree to refrain from sperm donation from check-in until 30 days beyond the conclusion of all study events.
* Male subjects must agree to the use of condoms with spermicide with sexual intercourse from 14 days prior to check-in until 30 days beyond the last dose of study drug.
* Resting heart rate ≥ 50 beats per minute (bpm)

Exclusion Criteria:

* History or presence of any clinically significant events, which in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Subjects with systolic blood pressure < 90 mmHg or diastolic blood pressure < 50 mmHg
* Male subjects with a QTcB > 450 msec
* Female subjects with a QTcB > 470 msec
* Subjects with pulmonary symptoms, history of exercise-induced asthma, asthma or chronic obstructive pulmonary disease (COPD)
* Use of any prescription drug within 1 month of starting the study
* Positive urine screen for alcohol or drugs at screening, unless the test is shown to be falsely positive on confirmation testing.
* Hemoglobin < 12g/dL
* Donation of blood or significant blood loss within 56 days prior to check in.
* Donation of plasma within 7 days prior check in.
* Participation in an investigational study within 30 days prior to check in.
* Positive screening test for HIV or Hepatitis B or C.
* A past history of cigarette smoking of > 10 pack-years or use of nicotine or nicotine-containing products 6 months prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Effects of two doses of FTY720 on lung and cardiac (heart) functions in healthy volunteers.

SECONDARY OUTCOMES:
Treatment initiation effect on heart rhythm.
Duration of dynamic effect on heart rate and rhythm.
Treatment initiation effect and duration of this effect on cardiac output and stroke volume.
Treatment initiation effect and the duration of this effect on pulmonary function with methacholine challenge.
Pharmacodynamic effect on absolute lymphocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States